CLINICAL TRIAL: NCT06950437
Title: Transcranial Magnetic Stimulation Guided by Personalized Brain Functional Sectors (pBFS) for Language Deficit Comorbid in Autism Spectrum Disorder Child: a Multi-center, Randomized, Sham-controlled Trial
Brief Title: pBFS Guided aiTBS Over Language Network for ASD Child
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Changping Tianhe Research Institute of Brain Science (Other)
Collaborators: Peking University Sixth Hospital (Other); Shanghai Yangzhi Rehabilitation Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NGASD002DMC_150
Record Dates: First submitted 2025-03-10; First posted 2025-04-30 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder; Language Delay
Keywords: ASD; language delay; aiTBS; precision neuromodulation
MeSH Terms: conditions — Autism Spectrum Disorder; Language Development Disorders | interventions — Speech Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active iTBS group (Experimental): active iTBS over SFG
  Interventions: Device: active iTBS; Behavioral: speech therapy
- Sham group (Sham Comparator): sham iTBS over SFG
  Interventions: Device: Sham iTBS; Behavioral: speech therapy

INTERVENTIONS:
Device: active iTBS — Participants will undergo three iTBS sessions per day, with 1800 pulses per session, over a 12-week period. Individualized targets will be generated using the pBFS technique.
  Arms: active iTBS group
Device: Sham iTBS — Participants will undergo three sham iTBS sessions per day, with 1800 pulses per session, over a 12-week period. Sham stimulation will be delivered through a sham coil with the identical appearance as real coil. Individualized targets will be generated using the pBFS technique.
  Arms: Sham group
Behavioral: speech therapy — Speech therapy will be delivered between iTBS/sham sessions. Two 30-minutes trainings every day.

SUMMARY:
The aim of this trial is to evaluate the efficacy and safety of precision neuromodulation in improving language ability in children with autism spectrum disorder (ASD) who also have language development delay. The neuromodulation will be delivered using the accelerated intermittent theta burst stimulation (aiTBS) protocol, targeting the language network in the left superior frontal gyrus (SFG), guided by personalized Brain Functional Sector (pBFS) technology.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is a neurodevelopmental disorder often accompanied by language delay. Emerging evidence indicates that Transcranial Magnetic Stimulation (TMS) has been effective in restoring language ability in post-stroke aphasia, but its efficacy in developmental language disorders remains unknown.

By leveraging the personalized Brain Functional Sector (pBFS) technique and task-free functional MRI scans, we can accurately locate the individual language function brain network. Considering the accessibility and comfort of neuromodulation, we will stimulate the language network node in the superior frontal gyrus (SFG) for 12 weeks.

In this study, participants meeting the inclusion and exclusion criteria will be randomly assigned to either the active or sham iTBS (intermittent theta burst stimulation) groups at a ratio of 2:1. The treatment protocol lasts for 12 weeks, with sessions held 5 days a week and 3 iTBS sessions over the SFG per day. The inter-session interval is set at 50 minutes, along with speech therapy. Clinical evaluations focusing on language and ASD symptoms will be conducted at baseline, after the 12-week treatment period, and at 24-week follow-up after the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Professionally diagnosed with ASD per DSM - 5 criteria.
2. Aged 3 - 6.5 years, either gender.
3. ADOS-2 results meet ASD standard cut - off.
4. SCQ score: ≥15 (age ≥ 4 years) or ≥11 (age < 4 years).
5. Co-existing language disorder not explaining ASD symptoms. No organic speech organ lesions. CNBS-R2016 and CLAS-TP language-related equivalent age > 18 months; any CLAS-TP dimension score < 6.
6. Mandarin is the daily communication language.
7. May have intellectual/global developmental delay not explaining ASD symptoms.
8. Guardians volunteer, can cooperate in treatment and sign informed consent.

Exclusion Criteria:

1. Identified genetic pathogenic factors; current/past comorbid severe disorders (ADHD, Tourette's, etc.).
2. Serious self-harm in the past year.
3. Severe sensory/motor disorders precluding cooperation.
4. History of epileptic seizures.
5. Serious organic diseases, especially brain related.
6. Contraindications for MRI/TMS (metal/implants).
7. Respiratory/circulatory diseases with sedation risk.
8. Illiterate guardians unable to handle informed consent/questionnaires.
9. Received neuromodulation in the past 3 months.
10. Currently in other clinical trials.
11. Deemed unfit by the researcher.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
CLAS-TP score change after treatment | Pre-treatment (baseline), post-treatment (12-week)
  The score changes of combined CLAS-TP (Child Language Assessment Scale - Test for Preschoolers) score at 12-week from baseline. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
CLAS-TP total score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  Higher scores mean a better outcome.
CLAS-TP subscale score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  For the story comprehension subscale, only participants who had non-zero point were included.
  Higher scores mean a better outcome.
WPPSI language score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  Higher scores mean a better outcome.
ADOS-2 SA score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  Higher scores mean a worse outcome.

OTHER OUTCOMES:
SCQ score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  Higher scores mean a worse outcome.
ATEC score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  Higher scores mean a worse outcome.
CBCL score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  Higher scores mean a worse outcome.
QoL score change from baseline to follow-up | Pre-treatment (baseline), post-treatment (12-week), follow-up (24-week)
  Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Sixth Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided